CLINICAL TRIAL: NCT03188445
Title: Intravenous Iron Isomaltoside Versus Oral Iron Supplementation for Treatment of Iron Deficiency in Pregnancy: a Randomised, Comparative, Open-label Trial
Brief Title: Intravenous Iron Isomaltoside Versus Oral Iron Supplementation for Treatment of Iron Deficiency in Pregnancy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-PREG-01
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Iron Deficiency Anemia of Pregnancy
MeSH Terms: interventions — iron isomaltoside 1000; ferrous fumarate; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV administration (Experimental): Iron isomaltoside (Monofer) Administered iv
  Interventions: Drug: Iron Isomaltoside 1000
- Oral administration (Active Comparator): Ferrous fumarate with ascorbic acid Administered oral
  Interventions: Drug: ferrous fumarate with ascorbic acid

INTERVENTIONS:
Drug: Iron Isomaltoside 1000 — Administered iv
  Arms: IV administration
Drug: ferrous fumarate with ascorbic acid — Oral administration
  Arms: Oral administration

SUMMARY:
Intravenous iron isomaltoside versus oral iron supplementation for treatment of iron deficiency in pregnancy

DETAILED DESCRIPTION:
Iron deficiency (ID) in pregnant women can cause iron deficiency anaemia (IDA). ID is defined by low iron stores, measured by a low level of s-ferritin. Iron is essential for the synthesis of haemoglobin (Hb). Anaemia is defined by a low Hb level (<11.0 g/dL in 1st trimester, <10.5 g/dL in 2nd, and <10.5 - 11.0 g/dL in 3rd trimesters).

In Danish pregnant women, who do not take iron supplementation approximately 50 % have ID and 21 % have IDA. According to WHO anaemia, defined as Hb <11.0 g/dL, regardless the cause is estimated to occur in 24 % of Danish pregnant women.

This trial is designed to evaluate and compare the effect of IV iron isomaltoside to a fixed dose of oral iron administered as tablet ferrous fumarate with ascorbic acid as correction of IDA in pregnant women after 4 weeks of standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥18 years
2. Pregnancy at GA 14+0 - 19+0
3. Ferritin <30 μg/L after 4 weeks of standard treatment in a clinical setting
4. Willingness to participate and attend all planned follow-up visits, and signing the in-formed consent form

Exclusion Criteria:

1. History of anaemia caused by e.g. thalassemia, hypersplenism or haemolytic anaemia (known haematologic disorder other than iron deficiency)
2. Iron overload or disturbances in utilisation of iron (e.g. haemochromatosis and haemosiderosis)
3. Drug hypersensitivity (i.e. previous hypersensitivity to IV iron)
4. Known hypersensitivity to any excipients in the investigational drug products
5. History of active asthma within the last 5 years
6. History of multiple allergies
7. Known decompensated liver cirrhosis or active hepatitis
8. Active acute or chronic infections (assessed by clinical judgement)
9. Rheumatoid arthritis with symptoms or signs of active inflammation
10. Treated with IV iron products or blood transfusion within 4 weeks prior to inclusion
11. Treated with erythropoietin (EPO) within 4 weeks prior to inclusion
12. Participation in any other interventional trial where the trial drug has not passed 5 half-lives prior to inclusion
13. Any other medical condition that, in the opinion of the Investigator, may cause the subject to be unsuitable for the completion of the trial or place the subject at potential risk from being in the trial
14. Meeting RBC-transfusion criteria (Hb ≤6.9 g/dL= 4.3 mmol/L with intolerable symptoms of anaemia like severe palpitations, severe dizziness, shortness of breath at rest or syncope or an Hb ≤6.4 g/dL (4.0 mmol/L) without intolerable symptoms of anaemia)
15. Multiple pregnancies
16. Inability to read and understand the Danish language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — A subject will be eligible for inclusion in the trial if she fulfils the following criteria:
  1. Women aged ≥18 years
  2. Pregnancy at GA 14+0 - 19+0
Enrollment: 201 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the achievement of an hemoglobin equal or above 11 g/dL | from baseline to 18 weeks after treatment

SECONDARY OUTCOMES:
Achievement of an hemoglobin equal to or above 11 g/dL | T=3 weeks, T=6 weeks, T=12 weeks, and T=18 weeks
Change in iron biomarkers | From baseline to T=3 weeks, T=6 weeks, T=12 weeks, and T=18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pharmacosmos A/S Clinical and Non-clinical Research, Study Director — Pharmacosmos A/S
Locations (1):
- Phamacosmos Investigational site, Hvidovre, Sjaeland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen R, Sommer VM, Pinborg A, Krebs L, Thomsen LL, Moos T, Holm C. Intravenous ferric derisomaltose versus oral iron for persistent iron deficient pregnant women: a randomised controlled trial. Arch Gynecol Obstet. 2023 Oct;308(4):1165-1173. doi: 10.1007/s00404-022-06768-x. Epub 2022 Sep 15. PMID 36107229
- [Derived] Markova V, Hansen R, Thomsen LL, Pinborg A, Moos T, Holm C. Intravenous iron isomaltoside versus oral iron supplementation for treatment of iron deficiency in pregnancy: protocol for a randomised, comparative, open-label trial. Trials. 2020 Aug 26;21(1):742. doi: 10.1186/s13063-020-04637-z. PMID 32843079